CLINICAL TRIAL: NCT00984139
Title: Long-term Persistence of Hepatitis B Antibodies and Immune Response to a Hepatitis B Vaccine Challenge in 12-13 Year Old Adolescents, Vaccinated in Infancy With GlaxoSmithKline (GSK) Biologicals' HBV Vaccine (Engerix™-B)
Brief Title: Persistence of Immunity Against Hepatitis B in 12-13 Year Old Adolescents After Infant Hepatitis B Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 112682
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2016-09

CONDITIONS: Hepatitis B
Keywords: persistence; HBV; Long-term; Engerix™-B Kinder; Hepatitis B; adolescent
MeSH Terms: conditions — Hepatitis B

ARMS (1):
- Engerix-B Group (Experimental): Subjects who were vaccinated with 3 doses of Engerix-B in infancy and who received a single challenge dose of Engerix-B , intramuscularly in the deltoid region of the non-dominant arm, at 12-13 years of age (Day 0).
  Interventions: Biological: Engerix™-B Kinder

INTERVENTIONS:
Biological: Engerix™-B Kinder — Intramuscular, one dose.
  Other Names: HBV vaccine; Engerix™-B

SUMMARY:
This phase IV open study will evaluate the persistence of humoral antibodies against hepatitis B as well as the immune response to a challenge dose of hepatitis B vaccine in adolescents aged 12-13 years, who received three consecutive doses of GSK Biologicals' recombinant hepatitis B vaccine (Engerix™-B) in infancy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Accepted representative (LAR(s)) can and will comply with the requirements of the protocol.
* A male or female of 12 to 13 years of age at the time of enrolment.
* With documented evidence of previous vaccination with three consecutive doses of Engerix-B in Germany: with the first two doses received by 9 months of age and the third dose received by 18 months of age.
* Written informed consent obtained from the parent(s) or LAR(s) of the subject at the time of enrolment.
* Written informed assent obtained from the subject in addition to the informed consent signed by the parent(s)/LAR(s).
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Females of childbearing potential at the time of study entry must have a negative pregnancy test prior to administration of the dose of vaccine and are required to be abstinent or to use adequate contraceptive precautions for one month prior to vaccination. Subjects are required to agree to continue such precautions for two months after vaccination.

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous hepatitis B booster vaccination since administration of the third dose of Engerix-B vaccine.
* History of hepatitis B disease.
* Hepatitis B vaccination at birth.
* Adolescents living in institutional care.
* Planned administration /administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before HBV vaccine challenge and ending 30 days after.
* Administration of immunoglobulins and/or any blood products within the three months preceding HBV vaccine challenge or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the HBV vaccine challenge..
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the challenge dose of study vaccine, or planned use during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Known hypersensitivity to any component of the HBV vaccine or evidence of hypersensitivity after previous immunisation with a vaccine containing the hepatitis B component.
* Acute disease and/or fever at the time of enrolment.

Ages: 12 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 306 (Actual)
Dates: Start 2009-10-12; Primary Completion 2010-04-07 (Actual); Study Completion 2010-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- Germany (21):
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Pforzheim, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Gilching, Bavaria
  - GSK Investigational Site, Kempten (Allgäu), Bavaria
  - GSK Investigational Site, Kirchheim, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Braunatal, Hesse
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Weimar, Thuringia
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Behre U, Bleckmann G, Crasta PD, Leyssen M, Messier M, Jacquet JM, Hardt K. Long-term anti-HBs antibody persistence and immune memory in children and adolescents who received routine childhood hepatitis B vaccination. Hum Vaccin Immunother. 2012 Jun;8(6):813-8. doi: 10.4161/hv.19898. Epub 2012 Apr 17. PMID 22508412
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 112682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Engerix-B Group
Started | 306
Completed | 306
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Engerix-B Group
Number analyzed (Participants) | 306
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.4 (0.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152
  Male | 154

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations as Measured by ELISA Equal to or Above Cut-off Value
Description: The cut-off value was defined as 100 milli-international units per milliliter (mIU/mL).
Time Frame: One month after the challenge dose (Month 1)
Population: The analysis was performed on the according-to-protocol (ATP) cohort of immunogenicity on all evaluable subjects who had received a challenge dose of Engerix-B and for whom data concerning immunogenicity outcome measures were available at the time point after the Engerix-B challenge dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Group
Number analyzed (Participants) | 284
Participants | 266

2. Primary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations as Measured by ChemiLuminescence ImmunoAssay (CLIA) Equal to or Above Cut-off Value.
Description: The cut-off value was defined as 100 milli-international units per milliliter (mIU/mL).
Time Frame: One month after the challenge dose (Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Group
Number analyzed (Participants) | 276
Participants | 257

3. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations as Measured by ELISA Equal to or Above Cut-off Values
Description: The cut-off values were defined as 3.3 mIU/mL, 10 mIU/mL and 100 mIU/mL.
  Note: the number of subjects with anti-HBs antibody concentrations equal to or above 100 mIU/mL on month post-challenge dose data are presented as a primary outcome measure.
Time Frame: Before (Day 0) and one month (Month 1) after the challenge dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Group
Number analyzed (Participants) | 284
Participants
  pre challenge dose 3.3 mIU/mL: number analyzed (Participants) | 282
  pre challenge dose 3.3 mIU/mL | 259
  post challenge dose 3.3 mIU/mL | 283
  pre challenge dose 10 mIU/mL: number analyzed (Participants) | 282
  pre challenge dose 10 mIU/mL | 220
  post challenge dose 10 mIU/mL | 281
  pre challenge dose 100 mIU/mL: number analyzed (Participants) | 282
  pre challenge dose 100 mIU/mL | 70

4. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations as Measured by CLIA Equal to or Above Cut-off Values
Description: The cut-off values were defined as 6.2 mIU/mL, 10 mIU/mL and 100 mIU/mL. Note: the number of subjects with anti-HBs antibody concentrations equal to or above 100 mIU/mL on month post-challenge dose data are presented as a primary outcome measure.
Time Frame: Before (Day 0) and one month (Month 1) after the challenge dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Group
Number analyzed (Participants) | 279
Participants
  pre challenge dose 6.2 mIU/mL | 201
  post challenge dose 6.2 mIU/mL: number analyzed (Participants) | 276
  post challenge dose 6.2 mIU/mL | 271
  pre challenge dose 10 mIU/mL | 181
  post challenge dose 10 mIU/mL: number analyzed (Participants) | 276
  post challenge dose 10 mIU/mL | 271
  pre challenge dose 100 mIU/mL | 67

5. Secondary Outcome: Number of Subjects With Solicited Local and General Symptoms
Description: Solicited local symptoms were pain, redness and swelling. Solicited general symptoms were fatigue, gastrointestinal symptoms, headache and fever.
  Fever was defined as axillary temperature greater than or equal to 37.5 degrees Celsius.
Time Frame: During the 4-day (Day 0-3) follow-up period following the challenge dose vaccination
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Group
Number analyzed (Participants) | 306
Participants
  pain | 104
  redness | 56
  swelling | 26
  fatigue | 63
  gastrointestinal symptoms | 14
  headache | 56
  fever | 9

6. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day (Day 0-30) follow-up period following the challenge dose vaccination
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Group
Number analyzed (Participants) | 306
Participants | 64

7. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: After the challenge dose of the vaccine (Day 0) up to the study end (Month 1)
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Group
Number analyzed (Participants) | 306
Participants | 0

8. Secondary Outcome: Number of Subjects With Anamnestic Response to the Challenge Dose as Measured by ELISA.
Description: Anamnestic response was defined as: - At least (i.e. greater than or equal to) a 4-fold rise in post-challenge vaccine dose anti-HBs antibody concentrations in subjects seropositive (i.e. with anti-HBs antibody concentration equal to or greater than 3.3 mIU/mL) at the pre-challenge dose time point. - Post-challenge dose anti-HBs antibody concentrations equal to or greater than 10 mIU/mL in subjects seronegative (i.e. with anti-HBs antibody concentrations less than 3.3 mIU/mL) at the pre-challenge dose time point.
Time Frame: One month after the challenge dose (Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Group
Number analyzed (Participants) | 282
Participants | 274

9. Secondary Outcome: Number of Subjects With Anamnestic Response to the Challenge Dose as Measured by CLIA.
Description: Anamnestic response was defined as: - At least (i.e. greater than or equal to) a 4-fold rise in post-challenge vaccine dose anti-HBs antibody concentrations in subjects seropositive (i.e. with anti-HBs antibody concentration ≥ 6.2 mIU/mL) at the pre-challenge dose time point. - Post-challenge dose anti-HBs antibody concentrations equal to or greater than 10 mIU/mL in subjects seronegative (i.e. with anti-HBs antibody concentrations < 6.2 mIU/mL) at the pre-challenge dose time point.
Time Frame: One month after the challenge dose (Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Group
Number analyzed (Participants) | 271
Participants | 267

ADVERSE EVENTS:
Arm/Group | Engerix-B Group
Serious Adverse Events (participants affected / at risk) | 0/306
Other Adverse Events (participants affected / at risk) | 170/306
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Engerix-B Group (N=306)
Pain (General disorders) | 104
Redness (General disorders) | 56
Swelling (General disorders) | 26
Fatigue (General disorders) | 63
Headache (General disorders) | 56

LIMITATIONS AND CAVEATS:
A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following complete retesting and reanalysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.